CLINICAL TRIAL: NCT06049212
Title: Phase 1 Trial of MK-2870 as Monotherapy and in Combination With Pembrolizumab ± Chemotherapy in Subjects With Advanced Solid Tumors
Brief Title: Sacituzumab Tirumotecan (MK-2870) as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors (MK-2870-008)
Acronym: TroFuse-008
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2870-008; jRCT2031230356 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer; Solid Tumors; Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Sacituzumab tirumotecan Monotherapy (Experimental): Participants receive single doses of sacituzumab tirumotecan monotherapy once every 2 weeks (Q2W).
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Supportive care measures
- Arm 2: Pembrolizumab + Sacituzumab tirumotecan Combination Therapy (Experimental): Participants receive sacituzumab tirumotecan Q2W in combination with pembrolizumab once every 6 weeks (Q6W).
  Interventions: Biological: Sacituzumab tirumotecan; Biological: Pembrolizumab; Drug: Supportive care measures

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — Sacituzumab tirumotecan injection powder for intravenous (IV) infusion.
  Other Names: SKB264; MK-2870
Biological: Pembrolizumab — Pembrolizumab solution for IV infusion.
  Other Names: MK-3475
  Arms: Arm 2: Pembrolizumab + Sacituzumab tirumotecan Combination Therapy
Drug: Supportive care measures — Participants are allowed to take supportive care measures at the discretion of the investigator. Prophylactic supportive care measures may include but are not limited to antiemetic agents, antidiarrheal agents, granulocyte and erythroid growth factors, and blood transfusions

SUMMARY:
This is a phase 1 trial of the safety, tolerability, and pharmacokinetics (PK) of sacituzumab tirumotecan monotherapy, and of sacituzumab tirumotecan in combination with pembrolizumab (MK-3475) or pembrolizumab + carboplatin, in Japanese participants with advanced solid tumors or treatment-naïve advanced or metastatic non-small cell lung cancer (NSCLC).

Per protocol amendment 04, Arm 3: Pembrolizumab/Carboplatin + sacituzumab tirumotecan Combination Therapy was discontinued, and subsequently all Arm 3 procedures, recruitment, and descriptions were removed.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1: Histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report and have received, or been intolerant to, all treatment known to confer clinical benefit.
* Arm 2: Have a histologically or cytologically confirmed diagnosis of advanced or metastatic NSCLC (Stage IIIB or IIIC disease and not candidates for surgical resection or definitive chemoradiation, or Stage IV NSCLC, AJCC Staging Manual, version 8).
* Arm 2: Confirmation that EGFR-, ALK-, or ROS1-directed therapy is not indicated as primary therapy
* Arm 2: Has tumor tissue that demonstrates PD-L1 TPS ≥ 50% as determined by PD-L1 IHC 22C3 pharmDx assay by local laboratory
* If capable of producing sperm, the participant agrees to the following during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention (100 days for sacituzumab tirumotecan and 90 days for carboplatin [no restriction for pembrolizumab]) AND agrees to refrain from donating sperm AND is either abstinent and agrees to remain abstinent or uses highly effective contraception
* For females (assigned at birth), is not pregnant or breastfeeding and ≥1 of the following applies: is not a participant of childbearing potential (POCBP) OR is a POCBP and uses highly effective contraception
* Arm 1: Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline
* Measurable disease by RECIST 1.1 as assessed by the local site investigator/radiology
* Archival tumor tissue sample or newly obtained core or incisional biopsy of a tumor lesion not previously irradiated has been provided
* Have a life expectancy of at least 3 months
* Have an ECOG performance status of 0 or 1 within 3 days before the start of study intervention

Exclusion Criteria:

* Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible
* Has Grade ≥2 peripheral neuropathy
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or severe corneal disease that prevents/delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of QTcF interval to >480 ms, and/or other serious cardiovascular and cerebrovascular diseases within the 6 months preceding study intervention
* Received prior treatment with a TROP2-targeted ADC
* Received prior treatment with a topoisomerase I-containing ADC
* Arm 1: Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis
* Arm 2: Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137)
* Arm 2: Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their advanced or metastatic NSCLC
* Arm 2: Has received radiation therapy to the lung that is >30 Gy within 6 months of the first dose of study intervention
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before allocation
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Requires treatment with a strong inhibitor or inducer of CYP3A4 at least 14 days before the first dose of study intervention and throughout the study
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Arm 2: Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Arm 2: Active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid)
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Known active CNS metastases and/or carcinomatous meningitis
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy
* History of HIV infection
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection
* History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorder
* A severe hypersensitivity reaction to treatment a monoclonal antibody/component of the study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicity (DLT) | Up to 21 days after each dose
  A DLT is defined as any of the following: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia or lymphopenia; any nonhematologic AE ≥Grade 3 in severity (with some exceptions); any Grade 3 or Grade 4 nonhematologic laboratory value (if certain criteria are met); febrile neutropenia Grade 3 or Grade 4; a prolonged delay (>2 weeks) in initiating sacituzumab tirumotecan second dose due to intervention-related toxicity; any intervention-related toxicity that causes the participant to discontinue intervention during DLT evaluation period; or any Grade 5 toxicity. All toxicities will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
Number of Participants Experiencing ≥1 Adverse Event (AE) | Up to ~32 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Discontinuing from Study Therapy due to AE | Up to ~32 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (AUC) of sacituzumab tirumotecan -Antibody-Drug Conjugate (sacituzumab tirumotecan ADC) | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The AUC of sacituzumab tirumotecan -ADC will be determined in participants from Arm 1.
Maximum Plasma Concentration (Cmax) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Cmax of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Minimum Plasma Concentration (Cmin) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Cmin of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Apparent terminal half-life (t½) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The t½ of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Time to Maximum Plasma Concentration (Tmax) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Tmax of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Clearance (CL) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The CL of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Volume of Distribution (Vz) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Vz of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Accumulation Ratio (Rac) of sacituzumab tirumotecan-ADC | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Rac of sacituzumab tirumotecan-ADC will be determined in participants from Arm 1.
Area Under the Plasma AUC of sacituzumab tirumotecan-Total Antibody (sacituzumab tirumotecan-TAB) | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The AUC of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
Cmax of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Cmax of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
Cmin of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Cmin of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
t½ of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The t½ of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
Tmax of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Tmax of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
CL of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The CL of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
Vz of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Vz of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
Rac of sacituzumab tirumotecan-TAB | Day 1: Preinfusion and 0.5, 2, 4, 8, 24, 48, and 72 hours postinfusion
  The Rac of sacituzumab tirumotecan-TAB will be determined in participants from Arm 1.
Cmax of sacituzumab tirumotecan-ADC Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Cmax of sacituzumab tirumotecan-ADC when coadministered with pembrolizumab will be determined in participants from Arm 2.
Cmin of sacituzumab tirumotecan-ADC Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Cmin of sacituzumab tirumotecan-ADC when coadministered with pembrolizumab will be determined in participants from Arm 2.
Rac of sacituzumab tirumotecan-ADC Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Rac of sacituzumab tirumotecan-ADC when coadministered with pembrolizumab will be determined in participants from Arm 2.
Cmax of sacituzumab tirumotecan-TAB Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Cmax of sacituzumab tirumotecan-TAB when coadministered with pembrolizumab will be determined in participants from Arm 2.
Cmin of sacituzumab tirumotecan-TAB Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Cmin of sacituzumab tirumotecan-TAB when coadministered with pembrolizumab will be determined in participants from Arm 2.
Rac of sacituzumab tirumotecan-TAB Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Rac of sacituzumab tirumotecan-TAB when coadministered with pembrolizumab will be determined in participants from Arm 2.
Cmax of KL610023 Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Cmax of KL610023 (free payload) when sacituzumab tirumotecan is coadministered with pembrolizumab will be determined in participants from Arm 2.
Rac of KL610023 Coadministered with Pembrolizumab | Cycle 1 and 2: Days 1 and 29 preinfusion and 0.5 hours postinfusion (each cycle is 29 days)
  The Rac of KL610023 (free payload) when sacituzumab tirumotecan is coadministered with pembrolizumab will be determined in participants from Arm 2.
Objective Response Rate (ORR) | Up to ~39 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Duration of Response (DOR) | Up to ~39 months
  DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause.
Incidence of Antidrug Antibodies (ADA) to sacituzumab tirumotecan | Up to ~32 months
  The incidence of ADA will be determined in participants from Arm 1 and Arm 2.
Incidence of Antidrug Antibodies (ADA) to pembrolizumab | Up to ~32 months
  The incidence of ADA will be determined in participants from Arm 2.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- Japan (7):
  - Aichi Cancer Center ( Site 0006), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0002), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0008), Matsuyama, Ehime
  - Kanagawa Cancer Center ( Site 0004), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 0007), Hirakata, Osaka
  - Shizuoka Cancer Center ( Site 0005), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 0001), Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com